CLINICAL TRIAL: NCT04584879
Title: Transdiagnostic Treatment Personalization: Prioritizing Therapy Components to Capitalize on Strengths or Compensate for Weaknesses
Brief Title: Transdiagnostic Treatment Personalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shannon E. Sauer-Zavala (Other)
Responsible Party: Sponsor-Investigator, Shannon E. Sauer-Zavala, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 53545
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Anxiety Disorders; Depressive Disorder; Post Traumatic Stress Disorder; Obsessive-Compulsive Disorder
Keywords: Unified Protocol; Cognitive Behavioral Therapy; Personalization
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Standard Group, Brief Intervention (Experimental): Participants in this group will receive 6 sessions of treatment in accordance with the standard, published Unified Protocol (UP) manual.
  Interventions: Behavioral: Standard UP Treatment
- Standard Group, Full Intervention (Experimental): Participants in this group will receive 12 sessions of treatment in accordance with the standard, published Unified Protocol (UP) manual.
  Interventions: Behavioral: Standard UP Treatment
- Capitalization Group, Brief Intervention (Experimental): Participants in this group will receive 6 sessions of treatment organized to prioritize skills that capitalize on patient strengths.
  Interventions: Behavioral: Capitalization UP Treatment
- Capitalization Group, Full Intervention (Experimental): Participants in this group will receive 12 sessions of treatment organized to prioritize skills that capitalize on patient strengths.
  Interventions: Behavioral: Capitalization UP Treatment
- Compensation Group, Brief Intervention (Experimental): Participants in this group will receive 6 sessions of treatment organized to prioritize skills that compensate for patient weaknesses.
  Interventions: Behavioral: Compensation UP Treatment
- Compensation Group, Full Intervention (Experimental): Participants in this group will receive 12 sessions of treatment organized to prioritize skills that compensate for patient weaknesses.
  Interventions: Behavioral: Compensation UP Treatment

INTERVENTIONS:
Behavioral: Standard UP Treatment — Participants will receive treatment modules sequenced in accordance with the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP; Barlow et al 2011; 2018).
  Arms: Standard Group, Brief Intervention; Standard Group, Full Intervention
Behavioral: Capitalization UP Treatment — Participants will receive Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) treatment modules organized to prioritize skills that capitalize on patient strengths.
  Arms: Capitalization Group, Brief Intervention; Capitalization Group, Full Intervention
Behavioral: Compensation UP Treatment — Participants will receive Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP) treatment modules organized to prioritize skills that compensate for patient weaknesses.
  Arms: Compensation Group, Brief Intervention; Compensation Group, Full Intervention

SUMMARY:
The primary purpose of this study is to explore whether the efficiency of treatment for anxiety and depressive disorders can be increased using two discrete strategies: personalized skill ordering and 2) treatment discontinuation based on proximal indicators of improvements. The present study will specifically use treatment components drawn from an evidence-based psychological intervention, the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UP). This intervention has strong empirical support for patients presenting with anxiety, depressive, and related disorders and contains therapeutic skills that are common in psychological interventions (e.g., psychoeducation, mindfulness training, cognitive restructuring, countering emotional avoidance, increasing interoceptive tolerance). This study will determine if prioritizing the order of treatment modules to capitalize on patient strengths or compensate for weakensses increases treatmen efficacy. Additionally, it will also identify under what conditions briefer treatment modules may be appropriate.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of at least one emotional disorder
* fluent in English
* medication stability

Exclusion Criteria:

* concurrent therapy
* psychological condition that would be better addressed by alternative treatments
* have received more than 5 sessions of cognitive behavioral therapy in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Severity | 12 weeks (baseline, week 6 and week 12)
  Clinical severity will be measured using the Diagnostic Interview for Anxiety, Mood, and Obsessive Compulsive and Related Neuropsychiatric Disorders (DIAMOND) dimensional clinician ratings. Scores range from 1-7; higher scores indicate greater severity.
Change in Anxiety Symptoms | 12 weeks (baseline, week 1, week, 2, week, 3.....week 12)
  Anxiety symptoms will be measured using the Overall Anxiety Severity and Interference Scale (OASIS). This is a self-report measure in which scores range from 0-20; higher scores indicate more severe anxiety symptoms.
Change in Depressive Symptoms | 12 weeks (baseline, week 1, week, 2, week, 3.....week 12)
  Depressive symptoms will be measured using the Overall Depression Severity and Interference Scale (ODSIS). This is a self-report measure in which scores range from 0-20; higher scores indicate more severe anxiety symptoms.
Change in Aversive Reactions to Emotions | 12 weeks (baseline, week 1, week, 2, week, 3.....week 12)
  Aversive reactions to emotions will be measured using the distress aversion subscale of the Multidimensional Experiential Avoidance Questionnaire (MEAQ). This is a self-report measure in which scores range from 13-78; higher scores indicate greater negative reactions to emotional experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Sauer-Zavala, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Southward MW, Terrill DR, Sauer-Zavala S. The effects of the Unified Protocol and Unified Protocol skills on loneliness in the COVID-19 pandemic. Depress Anxiety. 2022 Dec;39(12):913-921. doi: 10.1002/da.23297. Epub 2022 Nov 13. PMID 36372958